CLINICAL TRIAL: NCT07297342
Title: A Prospective Randomnised Controlled Trial Comparing Overall Patient Compliance in a Bariatric Surgical Pathway Using the Standard Versus a More Intensified and Interactive Version of the "Get Ready" Smartphone Application.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sint Dimpna Ziekenhuis Geel (Network)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ERP-2023-13530
Record Dates: First submitted 2025-09-23; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Obesity &Amp; Overweight; Hypertension; Obstructive Sleep Apnea (OSAS); Diabetes Mellitus ( Type 1 and Type 2)
Keywords: Get Ready; application; bariatric; compliance
MeSH Terms: conditions — Obesity; Overweight; Hypertension; Sleep Apnea, Obstructive; Diabetes Mellitus; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard GetReady application group (Placebo Comparator): Standard GetReady application group
  Interventions: Other: GetReady application
- Intensified GetReady application (Active Comparator): Intensified GetReady application
  Interventions: Other: Intensified GetReady application

INTERVENTIONS:
Other: GetReady application — Postoperative application usage
  Arms: Standard GetReady application group
Other: Intensified GetReady application — Postoperative application usage
  Arms: Intensified GetReady application

SUMMARY:
The aim of this study is to assess the impact of a newly intensified digital platform following bariatric surgery. This will be measured using several questionnaires. The following objectives will be evaluated: the exact amount of weight loss achieved preoperatively with the preparatory diet; the occurrence of dumping symptoms; the assessment of quality of life (QOL); and compliance with supplement intake.

By examining the impact of an enhanced digital platform, we aim to address critical questions regarding the effectiveness of improved patient support in the digital domain. Moreover, given the increasing prevalence of bariatric surgery as a therapeutic option for obesity, it is of utmost importance to identify strategies to optimize patient education and support through digital tools. This study not only contributes to the scientific understanding of digital support in bariatric care but also has important implications for the further development of the "Get Ready" application, ensuring that it remains at the forefront of providing comprehensive and patient-centered support in the evolving landscape of bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing bariatric surgery

Exclusion Criteria:

* Previous bariatric surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Weight | 3monts, 6 months, 12 months
  Overall weight, in kg's
Rand-36 Health Survey | 12months
  Health survey, score 0-100 with higher score indicating better health.
Bloodwork | 6 months and 12 months
  Deficiencys in blood results
Sigstad score | 3months, 6 months and 122 months
  classifying dumping symptoms, score >7 sugests dumping, score <-4 suggests other disease.

SECONDARY OUTCOMES:
N° of unplanned clinical visits | 12months
  N° of unplanned clinical visits

CONTACTS AND LOCATIONS:
Locations (1):
- Sint Dimpna ziekenhuis, Geel, Belgium